CLINICAL TRIAL: NCT04668235
Title: Evaluation of Safety and Clinical Efficacy of AZVUDINE in COVID-19 Patients (SARS-CoV-2 Infected): Phase III, Randomized, Double-blind, PLACEBO Controlled Trial
Brief Title: Study on Safety and Clinical Efficacy of AZVUDINE in COVID-19 Patients (SARS-CoV-2 Infected)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRH Pharmaceuticals Limited (Other)
Collaborators: GALZU INSTITUTE OF RESEARCH, TEACHING, SCIENCE AND APPLIED TECHNOLOGY, Brazil (Unknown); UNIVERSIDADE ESTADUAL DO NORTE FLUMINENSE (UENF), Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FNC IGZ-1
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: AZVUDINE; SARS-CoV-2; COVID-19; FNC
MeSH Terms: conditions — COVID-19 | interventions — azvudine; Cytosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm AZVUDINE (Experimental): Experimental:
  AZVUDINE 1mg tablet,
  Interventions:
  AZVUDINE 1mg tablet, 5 tablets QD + standard treatment for up to 14 days
  Interventions: Drug: AZVUDINE
- Arm Placebo (Placebo Comparator): Control:
  AZVUDINE placebo,
  Interventions:
  AZVUDINE placebo, 5 tablets QD + standard treatment for up to 14 days
  Interventions: Drug: AZVUDINE placebo

INTERVENTIONS:
Drug: AZVUDINE — 5 tablets QD + standard treatment for up to 14 days
  Other Names: AZVUDINE 1 mg tablets; FNC; 4-amino-1-((2R,3S,4R,5R)-5-azido-3-fluoro-4-hydroxy-5-(hydroxymethyl)tetrahydrofuran-2-yl)pyrimidine-2(1H)-one; 1-(4-Azido-2-deoxy-2-fluoro-beta-D- arabino Ribo-furanosyl) cytosine, FNC
  Arms: Arm AZVUDINE
Drug: AZVUDINE placebo — 5 tablets QD + standard treatment for up to 14 days
  Other Names: Placebo
  Arms: Arm Placebo

SUMMARY:
Estimated number of participants: 342 participants with COVID-19 Design: Phase III, single-center, randomized, double-blind, parallel, placebo-controlled clinical study.

In December 2021, there was a drop in the number of hospitalizations and the cases of COPD, tuberculosis and HIV associated with COVID-19, which are outside the inclusion criteria of this study. After the initial data of the study, there was a discussion with Anvisa and the size of the sample calculation was revised by amendment 4 (180 participants), and the methodology of statistical analysis for a new sample calculation was "a formula for sample calculation for superiority studies using proportions, according to the book do Chow et al (Chow, S.-C., Shao, J., Wang, H., &Lokhnygina, Y. Eds. 2017. Sample Size Calculations in Clinical Research: Third Edition, Chapman and Hall/CRC). Thus, Anvisa concluded that the adjustments are in accordance with the agency's guidelines, approving E4, which was later also approved by the Ethics Committee.

DETAILED DESCRIPTION:
Hypothesis:

AZVUDINE has therapeutic potential and safety profile for the treatment of patients infected with SARS-CoV-2.

Goals:

Primary objective • To assess the efficacy and safety of AZVUDINE (FNC) in relation to placebo, in patients infected with SARS-COV-2 in moderate to severe stage;

Secondary objective

• To evaluate the clinical outcome of the AZVUDINE group (FNC) compared to the placebo group in patients infected by SARS-COV-2 in moderate to severe stage;

Pharmaceutical form of the experimental medicine:

AZVUDINE 1 mg tablets

Comparators:

AZVUDINE placebo

Statistical planning:

The analyzes will be performed by FAS, PPS and SS and should be stratified by the severity of the disease (moderate, severe) and age (<60 years, ≥ 60 years), to assess the following parameters:

* Progression of the disease (moderate to severe, severe type);
* Negative viral load conversion rate;
* Time of negative conversion of viral load;
* Temperature recovery time;
* Time necessary to improve diarrhea, myalgia, fatigue, and other symptoms;
* Time to improve the pulmonary image;
* Frequency of supplemental oxygenation or non-invasive ventilation;
* Frequency of AEs;
* Mortality rate.

All statistical tests will be bilateral tests. If the P value is ≤0.05, it is considered that there is statistical significance between the difference in the tests.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 or over, regardless of gender;
2. Patients hospitalized in moderate to severe stages in line with the Ministry of Health classification;
3. Positive diagnosis for SARS-CoV-2 by molecular amplification of the virus in RT-PCR diagnosed from a respiratory sample (nasopharynx, oropharyngeal, lower respiratory tract [eg, sputum]) collected <96 hours before randomization;
4. Time of onset of symptoms and inclusion ≤ 14 days;
5. Internation within 48 hours after inclusion in the study;
6. Follow-up availability during the study period;
7. Voluntary membership to participate in the study and signing the Informed Consent Form.

Exclusion Criteria:

1. Patients known or suspected of being sensitive to AZVUDINE or excipients (inactive ingredients: microcrystalline cellulose, hydrated lactose, polyvinylpyrrolidone K30, croscarmellose sodium, magnesium stearate);
2. Patients diagnosed with pneumonia caused by other pathogens;
3. Patients with liver disease (total bilirubin ≥2 times above the normal limit, ALT / TGP and AST / TGO ≥5 times above the normal limit)
4. Patients with renal failure (glomerular filtration rate ≤60mL / min / 1.73 m2) or are receiving continuous renal replacement therapy, hemodialysis or peritoneal dialysis;
5. Individuals with malabsorption syndrome, or other conditions that affect gastrointestinal absorption, and circumstances in which patients need intravenous nutrition, or cannot take drugs orally or nasogastrically;
6. Pregnant or lactating women, or women with the potential to become pregnant during the study period and within 6 months after the end of administration;
7. Patients already included in other clinical trials;
8. Patient under treatment for HIV;
9. Patients being treated with other antivirals (eg lopinavir / ritonavir, remdesivir, umifenovir / arbidol, favipiravir, interferon-α)
10. Patients undergoing treatment with monoclonal antibodies (eg tocilizumab and sarilumab / kevzara);
11. Patients who are on a clinical treatment plan that includes the concomitant administration of any other experimental treatment or off-label use of drugs already on the market (eg hydroxychloroquine sulfate;
12. Patients who require invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) at the time of randomization;
13. Any clinically significant medical condition or medical history that, in the investigator's opinion, might discourage participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical improvement of AZVUDINE (FNC) in COVID-19 treatment | Day 1 to Day 15
  Rate of participants who reduced at least one level of the Clinical Progression Ordinal Scale category compared to the enrollment status (WHO, Jun/2020)

SECONDARY OUTCOMES:
Clinical cure outcome rate | Day 1 to Day 15
  Proportion of participants with clinical cure outcome during the study (viral RNA not detected and clinical conditions for discharge)
Recovery of body temperature | Day 1 to Day 28
  Time (days) for normalization of body temperature (below 37.6℃ axillary)
Clinical improvement of diarrhea, myalgia fatigue and other symptoms | Day 1 to Day 28
  Time (days) for clinical improvement of diarrhea, myalgia, fatigue, and other symptoms
Assessment of inflammatory biochemical markers (Reactive C Protein, erythrocyte sedimentation rate, and Procalcitonin) | Day 1 to Day 60
  Rate of change in biochemical markers of inflammatory function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
Assessment of immunological function biochemical markers (IL-6, IgG, IgM, IgA, and complement factor C3 and C4) | Day 1 to Day 60
  Rate of change in biochemical markers of immunological function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
Assessment of renal function biochemical markers (serum creatinine and calculated glomerular filtration rate) | Day 1 to Day 60
  Rate of change in biochemical markers of renal function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
Assessment of liver function biochemical markers (AST/TGO, ALT/TGP, ALP, GGT, BIL total, and direct BIL) | Day 1 to Day 60
  Rate of change in biochemical markers of hepatic function in relation to the physiological reference intervals between the AZVUDINA and PLACEBO groups.
Evaluation of time to negative conversion of SARS-CoV-2 viral load by RT-PCR | Day 1 to Day 28
  Time (days) to negative conversion of the SARS-CoV-2 viral load between AZVUDINE (FNC) and placebo group
Evaluation of the number of cycles for the detection of SARS-CoV-2 viral load by RT-PCR and application of the standard curve for calculating viral load | Day 1 to Day 15
  SARS-CoV-2 viral load determination by standard-curve method of quantification
Analysis of the relationship between the calculated viral load and the clinical evolution of the participants in the experimental group (FNC) and the PLACEBO group | Day 1 to Day 28
  Rating the relationship between viral load calculated and clinical outcomes of participants
Time for improvement of pulmonary condition by imaging exams during treatment | Day 1 to Day 28
  Time (days) for pulmonary image improvement of: (1) Ground glass opacity pattern, (2) mosaic paving, (3) alveolar consolidation, (4) reticular pattern / septal thickening, (5) opaque with inverted halo, (6) pleural / pericardial effusion, (7) fibrosis and / or (8) lymphadenomegaly.
Evaluation of pulmonary condition by imaging exams during treatment | Day 1 to Day 28
  Proportion of pulmonary image improvement of: (1) Ground glass opacity pattern, (2) mosaic paving, (3) alveolar consolidation, (4) reticular pattern / septal thickening, (5) opaque with inverted halo, (6) pleural / pericardial effusion, (7) fibrosis and / or (8) lymphadenomegaly.
Time for clinical improvement of respiratory signs and symptoms | Day 1 to Day 28
  Time (days) for improvement in respiratory signs and symptoms during treatment (pulmonary rales, cough, sputum, or sore throat)
Assessment of clinical improvement of respiratory signs and symptoms | Day 1 to Day 28
  Rate of improvement in respiratory signs and symptoms during treatment (pulmonary rales, cough, sputum, or sore throat)
Time for normalization of O2 saturation | Day 1 to Day 28
  Time (days) to normalize O2 saturation (above 95%) between AZVUDINE (FNC) and placebo group
Respiratory rate evaluation | Day 1 to Day 28
  Time (days) for respiratory rate normalization ≤24 rpm in room air
Frequency of supplemental oxygenation or non-invasive ventilation | Day 1 to Day 28
  Frequency of supplemental oxygenation or non-invasive ventilation
Frequency of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO | Day 1 to Day 28
  Frequency of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO
Proportion of moderate cases that progressed to severe cases | Day 1 to Day 28
  Proportion of moderate cases that progressed to severe cases requiring care in an intensive care unit
Assessment of hospitalization time | Day 1 to Day 28
  Length (days) of hospital stay
Evaluation of drug interaction events frequency | Day 1 to Day 28
  Frequency of drug interaction events
Evaluation of drug interaction events intensity | Day 1 to Day 28
  Intensity of drug interaction events (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Assessment of adverse events frequency | Day 1 to Day 28
  Frequency of adverse events
Assessment of adverse events intensity | Day 1 to Day 28
  Intensity of adverse events (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Assessment of unexpected adverse events frequency | Day 1 to Day 28
  Frequency of unexpected adverse events
Assessment of unexpected adverse events intensity | Day 1 to Day 28
  Intensity of unexpected adverse events (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Assessment of serious adverse events frequency | Day 1 to Day 28
  Frequency of serious adverse events
Assessment of serious adverse events intensity | Day 1 to Day 28
  Intensity of serious adverse events (1= Mild; 2= Moderate; 3= Severe; 4= Critical)
Overall mortality rate | Day 1 to Day 28
  Mortality rate during the study
Evaluation of the tolerability of azvudine in the 5 mg regimen orally QD up to 14 days | Day 1 to Day 28
  Treatment dropout rate due to AZVUDINE/Placebo intolerance.
Assessment of adherence of azvudine in the 5 mg regimen orally QD up to 14 days | Day 1 to Day 28
  Medication possession rate, to measure the proportion of administered dose episodes observed in relation to the expected number of doses, until treatment interruption.
Time of use of azvudine in the 5 mg regimen orally QD up to 14 days | Day 1 to Day 28
  Total time (days) of use of AZVUDINE / Placebo intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila P Figueiredo, MSc, Study Director — Galzu Institute
Locations (1):
- Santa Casa de Misericordia de Campos, Campos dos Goytacazes, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Souza SB, Cabral PGA, da Silva RM, Arruda RF, Cabral SPF, de Assis ALEM, Viana Junior AB, Degrave WMS, Moreira ADS, Silva CG, Chang J, Lei P. Phase III, randomized, double-blind, placebo-controlled clinical study: a study on the safety and clinical efficacy of AZVUDINE in moderate COVID-19 patients. Front Med (Lausanne). 2023 Oct 19;10:1215916. doi: 10.3389/fmed.2023.1215916. eCollection 2023. PMID 37928473